CLINICAL TRIAL: NCT00420368
Title: LCNI-6. A Single-centre Intervention Trial in Rural Malawi, Testing the Efficacy of Fortified Spread or Maize-soy Flour Supplementation to Alleviate Moderate Malnutrition Among 6-18 Month Old Children
Brief Title: Efficacy Trial on Alleviation of Infant Malnutrition With Fortified Spread or Maize-soy Flour Food Supplements
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Kamuzu University of Health Sciences (Other)
Responsible Party: Principal Investigator, Per Ashorn, Professor of International Health, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AF-109796-a
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Malnutrition
Keywords: Infant; Malnutrition; Sub-Saharan Africa; Treatment; Growth; Haemoglobin; Fortified spread; Food supplement
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: No food supplement
Dietary Supplement: Food supplement: fortified spread
Dietary Supplement: Food supplement: maize-soy flour

SUMMARY:
This study tests the hypothesis that moderately underweight but not severely wasted 6-17-month old infants receiving fortified spread or maize-soy flour as a food supplement for 12 weeks grow better during the supplementation than infants who do not get any food supplement.

DETAILED DESCRIPTION:
Childhood undernutrition is very common in rural Malawi, like in many other countries in Sub-Saharan Africa. Usually, undernutrition develops between 6 and 24 months of age. By two years of age, 30-50% of all children in rural Malawi are undernourished, predisposing them to subsequent morbidity, developmental delay and mortality. Urgent interventions are needed but the magnitude of the problem precludes a hospital-based management strategy. Therefore, emphasis must be on prevention and early home-based rehabilitation of children with mild-to-moderate malnutrition. However, the options for community based approaches are not as developed as those for institutional management of undernutrition.

The present study tests a recently developed micronutrient fortified spread, FS, which offers a potential solution to home based nutrition rehabilitation. The concept has previously been shown to work not only in therapeutic feeding of undernourished children in nutrition rehabilitation units in Malawi but also home based supplementation of undernourished children aged 42 to 60 months in Mangochi District, southern Malawi. In the present study the investigators will test the efficacy in growth promotion of this product when provided as a supplementary food to moderately underweight, but not wasted, infants (defined as WAZ <-2, WHM=>80%) between 6 and 18 months of age.

The study will be conducted in Lungwena area, Mangochi District, rural Malawi. A total of 189 6-15 -month old infants will be enrolled and randomised to three groups receiving different daily food supplements for 12 weeks. Children in group one (control group) will not receive any supplementation, children in group two will receive 300 g FS weekly (43 g / day) and children in group 3 will received 500 g of fortified maize/soy flour weekly (71 g / day). The food supplements will be delivered to the participant's home at weekly intervals.

All children will undergo medical and anthropometric examinations at 6-weekly intervals and disease symptoms monitoring every week. Dietary intake assessments will be conducted at 9 weeks after the onset of supplementation. A blood sample will be collected at the beginning and end of the study to measure blood haemoglobin and serum ferritin concentrations.

The impact of the dietary interventions will be primarily assessed by comparing weight gain in the three intervention groups. Secondary outcomes include length gain and changes in blood haemoglobin and serum ferritin concentration. The study will also produce descriptive data on morbidity and intake of foods during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent from at least one guardian
* age 6.00 months to 14.99 months
* weight-for-age <-2.0 Z scores
* availability during the period of the study.
* permanent resident Lungwena Health Centre catchment area

Exclusion Criteria:

* moderate or severe wasting (WHM<80% of the reference median)
* history of peanut allergy
* history of any serious allergic reaction to any substance, requiring emergency medical care
* history of anaphylaxis
* severe illness warranting hospital referral
* concurrent participation in another clinical trial with intervention to the child

Ages: 6 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 189
Dates: Start 2007-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Weight gain during the 12-week follow-up (in grams)

SECONDARY OUTCOMES:
Length gain during the 12-week follow-up (in centimetres)
Change in blood haemoglobin concentration during the study period (g/l)
Change in serum ferritin concentration during the study period (µg/l)
Change in anthropometric indices (WAZ, WHZ and HAZ)
Proportion developing moderate or severe wasting during the intervention (WHM<80% of the reference median)
Change in mid-upper arm and head circumference

CONTACTS AND LOCATIONS:
Overall Officials: Per Ashorn, MD, PhD, Study Director — University of Tampere, Medical School, Finland; Kenneth Maleta, MBBS, PhD, Principal Investigator — University of Malawi, College of Medicine, Department of Community Health
Locations (1):
- College of Medicine, University of Malawi, Mangochi, Mangochi District, Malawi

REFERENCES:
- [Result] Thakwalakwa C, Ashorn P, Phuka J, Cheung YB, Briend A, Puumalainen T, Maleta K. A lipid-based nutrient supplement but not corn-soy blend modestly increases weight gain among 6- to 18-month-old moderately underweight children in rural Malawi. J Nutr. 2010 Nov;140(11):2008-13. doi: 10.3945/jn.110.122499. Epub 2010 Sep 22. PMID 20861218
- See also: College of Medicine home page — http://www.medcol.mw/